CLINICAL TRIAL: NCT01202565
Title: Effectiveness of Adalimumab (Humira) in the Treatment of Scalp and Nail Affection in Patients With Moderate to Severe Plaque Psoriasis in Routine Clinical Practice
Brief Title: Effectiveness of Adalimumab (HUMIRA®) in the Treatment of Scalp and Nail Affection in Patients With Moderate to Severe Plaque Psoriasis in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-165
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Post-marketing observational study (PMOS) Protocol; Moderate to Severe Plaque Psoriasis; Treatment of Scalp and Nail Affection; Effectiveness of Adalimumab (HUMIRA®)

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: Participants with moderate to severe plaque psoriasis received adalimumab (Humira®) therapy according to the local product label and prescription/reimbursement guidelines.

SUMMARY:
There is clearly a need for further data on the efficacy of biologic agents in the treatment of nail and scalp psoriasis, especially in the routine clinical setting. A few case reports can be found, but no published data exists from non-interventional studies, such as post-marketing observational studies (PMOS) that reflect routine clinical practice.

The aim of this PMOS is to evaluate the long-term (12-month) efficacy of adalimumab in the treatment of nail and scalp psoriatic lesions in routine dermatologic practice.

DETAILED DESCRIPTION:
This is post-marketing observational study (PMOS) in which HUMIRA® is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication, and following the local prescription and/or reimbursement guidance.

Follow-up visits are not strictly scheduled, but rather left to the judgment of each investigator within the 12-month study period for each participant. Five visits are indicated within the 12-month observational period: Baseline and follow-up at 3 months, 6 months, 9 months and at 12 months (Study End).

As nails are not included in the general measures of disease severity (such as Psoriasis Area and Severity Index [PASI]), the Nail Psoriasis Severity Index (NAPSI) will be used to assign a score of nail psoriasis. The scalp, though being involved in the general measures of disease severity (e.g. PASI), represents only 4-5% of the body surface and is therefore poorly represented. Psoriasis Scalp Severity Index (PSSI) will be used to quantify the intensity of scalp psoriasis and its changes during the study. The association between general skin and localized nail and scalp, and changes in quality of life in response to adalimumab therapy will also be examined.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled in this PMOS if they fulfill all of the below criteria:

1. Patients with moderate to severe plaque psoriasis eligible for Humira therapy according to the local product label and prescription/reimbursement guidelines
2. Have significant psoriatic nail affection (total Nail Psoriasis Severity Index NAPSI score of hands and feet ≥ 10) and/or significant psoriatic scalp affection (Psoriasis Scalp Severity Index PSSI score ≥ 10)
3. Adult (≥18 years of age)
4. Have negative result of tuberculosis (TB) screening test or TB prophylaxis as per local guidelines
5. Willing to provide informed consent if requested by the local law regulations

Exclusion Criteria:

Patients fulfilling any of the below exclusion criteria will not be eligible for this PMOS:

1. Meet contraindications as outlined in the latest version of the local Summary of Product Characteristics (SmPC)
2. Participate in another clinical/observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Per this PMOS protocol, the study population will consists of adult patients with moderate to severe plaque psoriasis who have failed to respond to, have a contraindication to, or are intolerant of other systemic therapies including cyclosporine, methotrexate or PUVA (photochemotherapy combining psoralen with ultraviolet A treatment), and exhibit a significant psoriatic affection of the scalp and/or nails.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaka Brumen, Study Director — AbbVie
Locations (73):
- Czechia (8):
  - Site Reference ID/Investigator# 63776, Chotoviny
  - Site Reference ID/Investigator# 58083, Jihlava
  - Site Reference ID/Investigator# 56762, Klimkovice
  - Site Reference ID/Investigator# 56763, Klimkovice
  - Site Reference ID/Investigator# 30742, Kostelec nad Ohří
  - Site Reference ID/Investigator# 54503, Prague
  - Site Reference ID/Investigator# 56542, Prague
  - Site Reference ID/Investigator# 58084, Prague
- Estonia (4):
  - Site Reference ID/Investigator# 57562, Tallinn
  - Site Reference ID/Investigator# 57563, Tallinn
  - Site Reference ID/Investigator# 57564, Tallinn
  - Site Reference ID/Investigator# 57567, Tartu
- Hungary (15):
  - Site Reference ID/Investigator# 30743, Budapest
  - Site Reference ID/Investigator# 42506, Debrecen
  - Site Reference ID/Investigator# 42507, Debrecen
  - Site Reference ID/Investigator# 42508, Debrecen
  - Site Reference ID/Investigator# 42509, Debrecen
  - Site Reference ID/Investigator# 42510, Debrecen
  - Site Reference ID/Investigator# 42514, Kaposvár
  - Site Reference ID/Investigator# 42515, Kecskemét
  - Site Reference ID/Investigator# 42516, Miskolc
  - Site Reference ID/Investigator# 42511, Pécs
  - Site Reference ID/Investigator# 42512, Pécs
  - Site Reference ID/Investigator# 42513, Pécs
  - Site Reference ID/Investigator# 44854, Pécs
  - Site Reference ID/Investigator# 42502, Szeged
  - Site Reference ID/Investigator# 42517, Szombathely
- Israel (5):
  - Site Reference ID/Investigator# 30744, Afula
  - Site Reference ID/Investigator# 49888, Jerusalem
  - Site Reference ID/Investigator# 49886, Petach Tiqwa
  - Site Reference ID/Investigator# 49887, Ramat Gan
  - Site Reference ID/Investigator# 51783, Tel Aviv
- Romania (26):
  - Site Reference ID/Investigator# 46184, Alexandria
  - Site Reference ID/Investigator# 44580, Bucharest
  - Site Reference ID/Investigator# 44572, Bucharest
  - Site Reference ID/Investigator# 44575, Bucharest
  - Site Reference ID/Investigator# 44576, Bucharest
  - Site Reference ID/Investigator# 46185, Bucharest
  - Site Reference ID/Investigator# 44563, Bucharest
  - Site Reference ID/Investigator# 44564, Bucharest
  - Site Reference ID/Investigator# 44566, Bucharest
  - Site Reference ID/Investigator# 44567, Bucharest
  - Site Reference ID/Investigator# 44569, Bucharest
  - Site Reference ID/Investigator# 44571, Bucharest
  - Site Reference ID/Investigator# 30745, Cluj-Napoca
  - Site Reference ID/Investigator# 44561, Constanța
  - Site Reference ID/Investigator# 44562, Constanța
  - Site Reference ID/Investigator# 44557, Craiova
  - Site Reference ID/Investigator# 44558, Craiova
  - Site Reference ID/Investigator# 44559, Craiova
  - Site Reference ID/Investigator# 44560, Craiova
  - Site Reference ID/Investigator# 44547, Iași
  - Site Reference ID/Investigator# 44548, Iași
  - Site Reference ID/Investigator# 44549, Iași
  - Site Reference ID/Investigator# 46183, Oradea
  - Site Reference ID/Investigator# 44555, Ploieşti
  - Site Reference ID/Investigator# 44554, Reghin
  - Site Reference ID/Investigator# 44550, Târgu Mureş
- Slovakia (5):
  - Site Reference ID/Investigator# 30746, Banská Bystrica
  - Site Reference ID/Investigator# 42521, Bratislava
  - Site Reference ID/Investigator# 42519, Košice
  - Site Reference ID/Investigator# 42522, Martin
  - Site Reference ID/Investigator# 42518, Prešov
- Slovenia (4):
  - Site Reference ID/Investigator# 30747, Ljubljana
  - Site Reference ID/Investigator# 44544, Ljubljana
  - Site Reference ID/Investigator# 44542, Maribor
  - Site Reference ID/Investigator# 47702, Sežana
- Ukraine (6):
  - Site Reference ID/Investigator# 64524, Donetsk
  - Site Reference ID/Investigator# 66642, Donetsk
  - Site Reference ID/Investigator# 62304, Kharkiv
  - Site Reference ID/Investigator# 56699, Kiev
  - Site Reference ID/Investigator# 55443, Lviv
  - Site Reference ID/Investigator# 70493, Lviv

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Slovenia, Hungary, Slovakia, Romania, Israel, Czech Republic, Ukraine and Estonia.
Pre-assignment Details: Reasons for study discontinuation were not systematically collected. Five participants were lost to follow-up after the Baseline visit and had no entries regarding treatment with adalimumab and were excluded from the full analysis set (FAS) which finally comprises 501 participants.
Period: Overall Study
Arm/Group | Adalimumab
Started | 506
Full Analysis Set | 501 (Participants with a signed informed consent and any available data regarding adalimumab treatment.)
Completed | 439 (Indicates participants who completed the Month 12 visit)
Not Completed | 67

BASELINE CHARACTERISTICS:
Population: Full analysis set, which included participants with a signed informed consent and with any available data regarding treatment with adalimumab.
Arm/Group | Adalimumab
Number analyzed (Participants) | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 314
Nail Psoriasis Severity Index (NAPSI) Score [Mean (Standard Deviation); unit: units on a scale] — The NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The sum of these two scores is the total score for that nail. In this study the 2 most affected nails on either hands or feet were evaluated for a score ranging from 0 (no nail psoriasis) to 16 (psoriasis in 4/4 nail quadrants). Data are reported for the Nail Psoriasis Set (NPS), which includes participants with a Baseline NAPSI value ≥ 10 (157 participants).
  units on a scale | 13.0 (2.1)
Psoriasis Scalp Severity Index (PSSI) Score [Mean (Standard Deviation); unit: units on a scale] — PSSI consists of an assessment of scalp area involved and an assessment of the 3 clinical symptoms erythema, induration and desquamation. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). The total score ranges from 0 (best) to 72 (worst) and is derived from the sum of symptom scores multiplied by the score of involved scalp area. Data are reported for the Scalp Psoriasis Set (SPS), which includes participants with a Baseline PSSI value ≥ 10 (404 participants).
  units on a scale | 26.8 (14.1)
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. PASI data were missing for 2 participants at Baseline.
  units on a scale | 22.0 (9.7)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 (best) to 30 (worst). Baseline DLQI data were available for 459 participants.
  units on a scale | 20.0 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Nail Psoriasis Severity Index (NAPSI) to Month 12
Description: NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The sum of these two scores is the total score for that nail. Nail matrix psoriasis consists of any of the following: pitting, leukonychia, red spots in the lunula, or nail plate crumbling. Nail bed psoriasis is the presence or absence of onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration or nail bed hyperkeratosis. Scoring for each is based on the following scale:
  * 0 = none;
  * 1 = present in 1/4 nail quadrants;
  * 2 = present in 2/4 nail quadrants;
  * 3 = present in 3/4 nail quadrants;
  * 4 = present in 4/4 nail quadrants.
  The 2 most affected nails on either hands or feet were evaluated and summed for a score ranging from 0 (no nail psoriasis) to 16 (psoriasis in 4/4 nail quadrants).
  Change from Baseline is presented as a percentage of the Baseline value, calculated as: Month 12 value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 12
Population: Nail Psoriasis set, which includes participants with a Baseline NAPSI score ≥ 10. Only participants with a Baseline and at least one post-baseline value are included. Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 156
percent change | -74.6 (26.9)

2. Primary Outcome: Percent Change From Baseline in Psoriasis Scalp Severity Index (PSSI) to Month 12
Description: The PSSI consists of two parts: an assessment of scalp area involved and an assessment of the 3 clinical symptoms erythema, induration and desquamation. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). The composite score ranges from 0 (best) to 72 (worst) and is derived from the sum of symptom scores multiplied by the score of involved scalp area.
  Change from Baseline is presented as a percentage of the Baseline value: Month 12 value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 12
Population: Scalp Psoriasis Set (SPS), which includes participants with a Baseline PSSI ≥ 10. Only participants with a Baseline and at least one post-baseline value are included. Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 402
percent change | -89.7 (30.0)

3. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI)
Description: NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The sum of these two scores is the total score for that nail. Nail matrix psoriasis consists of any of the following: pitting, leukonychia, red spots in the lunula, or nail plate crumbling. Nail bed psoriasis is the presence or absence of onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration or nail bed hyperkeratosis. Scoring for each is based on the following scale:
  * 0 = none;
  * 1 = present in 1/4 nail quadrants;
  * 2 = present in 2/4 nail quadrants;
  * 3 = present in 3/4 nail quadrants;
  * 4 = present in 4/4 nail quadrants.
  The 2 most affected nails on either hands or feet were evaluated and summed for a score ranging from 0 (no nail psoriasis) to 16 (psoriasis in 4/4 nail quadrants).
  A negative change from Baseline indicates improvement.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: Nail Psoriasis Set; the analysis was based on all available data. Last observation carried forward (LOCF) was also used for the Month 12 time point. The number of participants included in the analysis at each time point is indicated by "N."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 157
units on a scale
  Month 3 (N=154) | -4.6 (3.0)
  Month 6 (N=144) | -7.6 (3.2)
  Month 9 (N=136) | -9.1 (3.5)
  Month 12 (N=125) | -10.5 (3.1)
  Month 12-LOCF (N=156) | -9.6 (3.7)

4. Secondary Outcome: Percentage of Participants Achieving a Good Clinical Response on Nail Psoriasis
Description: Good clinical response on nails is defined as ≥ 50% improvement from Baseline in total NAPSI score.
  The NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The sum of these two scores is the total score for that nail. Nail matrix psoriasis consists of any of the following: pitting, leukonychia, red spots in the lunula, or nail plate crumbling. Nail bed psoriasis is the presence or absence of onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration or nail bed hyperkeratosis. Scoring for each is based on the following scale:
  * 0 = none;
  * 1 = present in 1/4 nail quadrants;
  * 2 = present in 2/4 nail quadrants;
  * 3 = present in 3/4 nail quadrants;
  * 4 = present in 4/4 nail quadrants.
  The 2 most affected nails on either hands or feet were evaluated and summed for a score ranging from 0 (no nail psoriasis) to 16 (psoriasis in 4/4 nail quadrants).
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 157
percentage of participants
  Month 3 (N=154) | 33.1
  Month 6 (N=144) | 68.1
  Month 9 (N=136) | 85.3
  Month 12 (N=125) | 90.4
  Month 12-LOCF (N=156) | 84.0

5. Secondary Outcome: Percentage of Participants Achieving Complete Clearing of Nails
Description: Complete clearing of nails is defined as a total NAPSI score of zero.
  The NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The sum of these two scores is the total score for that nail. Nail matrix psoriasis consists of any of the following: pitting, leukonychia, red spots in the lunula, or nail plate crumbling. Nail bed psoriasis is the presence or absence of onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration or nail bed hyperkeratosis. Scoring for each is based on the following scale:
  * 0 = none;
  * 1 = present in 1/4 nail quadrants;
  * 2 = present in 2/4 nail quadrants;
  * 3 = present in 3/4 nail quadrants;
  * 4 = present in 4/4 nail quadrants.
  The 2 most affected nails on either hands or feet were evaluated and summed for a score ranging from 0 (no nail psoriasis) to 16 (psoriasis in 4/4 nail quadrants).
Time Frame: Months 3, 6, 9, and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 157
percentage of participants
  Month 3 (N=154) | 1.9
  Month 6 (N=144) | 11.8
  Month 9 (N=136) | 22.1
  Month 12 (N=125) | 40.0
  Month 12-LOCF (N=156) | 33.3

6. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI)
Description: The PSSI consists of two parts: an assessment of scalp area involved and an assessment of the 3 clinical symptoms erythema, induration and desquamation. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). The composite score ranges from 0 (best) to 72 (worst) and is derived from the sum of symptom scores multiplied by the score of involved scalp area. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: Scalp Psoriasis Set; the analysis was based on all available data. Last observation carried forward (LOCF) was also used for the Month 12 time point. The number of participants included in the analysis at each time point is indicated by "N."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 404
units on a scale
  Month 3 (N=400) | -17.2 (11.6)
  Month 6 (N=377) | -22.2 (12.7)
  Month 9 (N=365) | -24.2 (14.0)
  Month 12 (N=346) | -25.8 (14.5)
  Month 12-LOCF (N=402) | -24.3 (15.1)

7. Secondary Outcome: Percentage of Participants Achieving Good Clinical Response on Scalp
Description: Good clinical response on scalp is defined as a ≥ 50% improvement from Baseline in PSSI score.
  The PSSI consists of two parts: an assessment of scalp area involved and an assessment of the 3 clinical symptoms erythema, induration and desquamation. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). The composite score ranges from 0 (best) to 72 (worst) and is derived from the sum of symptom scores multiplied by the score of involved scalp area.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 404
percentage of participants
  Month 3 (N=400) | 67.0
  Month 6 (N=377) | 92.8
  Month 9 (N=365) | 97.5
  Month 12 (N=346) | 98.3
  Month 12-LOCF (N=402) | 93.8

8. Secondary Outcome: Percentage of Participants Achieving Complete Clearing of Scalp
Description: Complete clearing on scalp is defined as a PSSI score of zero. The PSSI consists of two parts: an assessment of scalp area involved and an assessment of the 3 clinical symptoms erythema, induration and desquamation. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). The composite score ranges from 0 (best) to 72 (worst) and is derived from the sum of symptom scores multiplied by the score of involved scalp area.
Time Frame: Months 3, 6, 9, and 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 404
percentage of participants
  Month 3 (N=400) | 27.0
  Month 6 (N=377) | 39.5
  Month 9 (N=365) | 47.9
  Month 12 (N=346) | 71.7
  Month 12-LOCF (N=402) | 66.7

9. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Change from Baseline is presented as a percentage of the Baseline value: Month 12 value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 12
Population: Full analysis Set. Only participants with a Baseline and at least one post-baseline value are included. Last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 495
percent change | -83.3 (36.0)

10. Secondary Outcome: Change From Baseline in PASI Score
Description: The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: Full Analysis Set with Baseline PASI score; the analysis was based on all available data. Last observation carried forward (LOCF) was also used for the Month 12 time point. The number of participants included in the analysis at each time point is indicated by "N."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 499
units on a scale
  Month 3 (N=490) | -14.5 (10.1)
  Month 6 (N=468) | -17.9 (10.2)
  Month 9 (N=449) | -19.6 (10.1)
  Month 12 (N=429) | -20.6 (9.9)
  Month 12-LOCF (N=495) | -19.1 (11.0)

11. Secondary Outcome: Percentage of Participants Achieving a PASI 90 Response
Description: The percentage of participants with a ≥ 90% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline.
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 499
percentage of participants
  Month 3 (N=490) | 25.1
  Month 6 (N=468) | 38.0
  Month 9 (N=449) | 51.4
  Month 12 (N=429) | 72.0
  Month 12-LOCF (N=495) | 65.3

12. Secondary Outcome: Percentage of Participants Achieving a PASI 75 Response
Description: The percentage of participants with a ≥ 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline.
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 499
percentage of participants
  Month 3 (N=490) | 43.5
  Month 6 (N=468) | 66.7
  Month 9 (N=449) | 84.6
  Month 12 (N=429) | 91.8
  Month 12-LOCF (N=495) | 84.0

13. Secondary Outcome: Percentage of Participants Achieving a PASI 50 Response
Description: The percentage of participants with a ≥ 50% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline.
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 499
percentage of participants
  Month 3 (N=490) | 69.2
  Month 6 (N= 468) | 92.5
  Month 9 (N=449) | 95.5
  Month 12 (N= 429) | 97.2
  Month 12-LOCF (N=495) | 91.1

14. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. Change from Baseline is presented as a percentage of the Baseline value: Month 12 value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 452
percent change | -83.6 (41.8)

15. Secondary Outcome: Change From Baseline in DLQI Score
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: Full Analysis Set with Baseline DLQI score; the analysis was based on all available data. Last observation carried forward (LOCF) was also used for the Month 12 time point. The number of participants included in the analysis at each time point is indicated by "N."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 459
units on a scale
  Month 3 (N=448) | -12.6 (7.1)
  Month 6 (N=426) | -16.1 (7.2)
  Month 9 (N=415) | -17.9 (7.0)
  Month 12 (N=396) | -18.9 (6.9)
  Month 12-LOCF (N=453) | -17.4 (8.4)

16. Secondary Outcome: Associations Between General Improvement in Psoriasis With Improvement in Nail Psoriasis
Description: Associations between general improvement in psoriasis, measured by percentage change of PASI, and the improvement of nail psoriasis at the same time, measured by percentage improvement of the NAPSI, were evaluated by means of Spearman's rank correlation coefficient. Generally, correlation coefficients below 0.2 are considered as no or only weak association, between 0.2 and 0.5 as moderate association, between 0.5 and 0.8 as strong association and above 0.8 as very strong associations.
Time Frame: Baseline and Month 12
Population: Nail Psoriasis Set; participants with both NAPSI and PASI data available. LOCF was used.
Measure: Number; unit: correlation coefficient
Arm/Group | Adalimumab
Number analyzed (Participants) | 155
correlation coefficient | 0.61

17. Secondary Outcome: Associations Between General Improvement in Psoriasis With Improvement in Scalp Psoriasis
Description: Associations between general improvement in psoriasis, measured by percentage change of PASI, and the improvement of scalp psoriasis at the same time, measured by percentage improvement of the PSSI, were evaluated by means of Spearman's rank correlation coefficient. Generally, correlation coefficients below 0.2 are considered as no or only weak association, between 0.2 and 0.5 as moderate association, between 0.5 and 0.8 as strong association and above 0.8 as very strong associations.
Time Frame: Baseline and Month 12
Population: Scalp Psoriasis Set; participants with both PSSI and PASI data available. LOCF was used.
Measure: Number; unit: correlation coefficient
Arm/Group | Adalimumab
Number analyzed (Participants) | 399
correlation coefficient | 0.65

18. Secondary Outcome: Associations Between Improvement in Quality of Life With Improvement in Nail Psoriasis
Description: Associations between general improvement in quality of life, measured by percentage change of DLQI, and the improvement of nail psoriasis at the same time, measured by percentage improvement of the NAPSI, were evaluated by means of Spearman's rank correlation coefficient. Generally, correlation coefficients below 0.2 are considered as no or only weak association, between 0.2 and 0.5 as moderate association, between 0.5 and 0.8 as strong association and above 0.8 as very strong associations.
Time Frame: Baseline and Month 12
Population: Nail Psoriasis Set; participants with both NAPSI and DLQI data available. LOCF was used.
Measure: Number; unit: correlation coefficient
Arm/Group | Adalimumab
Number analyzed (Participants) | 139
correlation coefficient | 0.60

19. Secondary Outcome: Associations Between Improvement in Quality of Life With Improvement in Scalp Psoriasis
Description: Associations between general improvement in quality of life, measured by percentage change of DLQI, and the improvement of scalp psoriasis at the same time, measured by percentage improvement of the PSSI, were evaluated by means of Spearman's rank correlation coefficient. Generally, correlation coefficients below 0.2 are considered as no or only weak association, between 0.2 and 0.5 as moderate association, between 0.5 and 0.8 as strong association and above 0.8 as very strong associations.
Time Frame: Baseline and Month 12
Population: Scalp Psoriasis Set; participants with both PSSI and DLQI data available. LOCF was used.
Measure: Number; unit: correlation coefficient
Arm/Group | Adalimumab
Number analyzed (Participants) | 376
correlation coefficient | 0.59

20. Secondary Outcome: Associations Between General Improvement in Psoriasis With Improvement in Quality of Life
Description: Associations between general improvement in quality of life, measured by percentage change of DLQI, and general improvement in psoriasis at the same time, measured by percentage improvement of the PASI, were evaluated by means of Spearman's rank correlation coefficient. Generally, correlation coefficients below 0.2 are considered as no or only weak association, between 0.2 and 0.5 as moderate association, between 0.5 and 0.8 as strong association and above 0.8 as very strong associations.
Time Frame: Baseline and Month 12
Population: Full Analysis Set; participants with both PASI and DLQI data available. LOCF was used.
Measure: Number; unit: correlation coefficient
Arm/Group | Adalimumab
Number analyzed (Participants) | 450
correlation coefficient | 0.78

ADVERSE EVENTS:
Time Frame: 12 months
Description: The analysis of adverse events was performed for the full analysis set
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 5/501
Other Adverse Events (participants affected / at risk) | 19/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=501)
Death (General disorders) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Polyneuropathy alcoholic (Nervous system disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=501)
Psoriasis (Skin and subcutaneous tissue disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.